CLINICAL TRIAL: NCT03191474
Title: CCTG 602: Linkage of Transgender Individuals to PrEP, A Multicenter Trial of the California Collaborative Treatment Group (CCTG)
Brief Title: Linkage of Transgender Individuals to PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Los Angeles LGBT Center (Other)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCTG 602
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: HIV Seronegativity; Linkage
Keywords: PrEP; Pre-exposure Prophylaxis; Truvada; Client-centered case management; Transgender; Gender non-conforming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (No Intervention): Participants will receive standard of care HIV risk assessment, PrEP education, and an appointment for a PrEP evaluation visit at an affiliated clinic.
- T-POWr Intervention Arm (Experimental): Participants will receive the same HIV risk assessment, PrEP education, and appointment for a PrEP evaluation visit as the Control Arm. Participants in the Intervention Arm will also receive a thorough client-centered case management evaluation that will assess needs including access to health insurance, general health care, assessment of current hormone administration, housing, mental health care, domestic violence care, substance use treatment, and other services.
  Interventions: Behavioral: T-POWr Intervention

INTERVENTIONS:
Behavioral: T-POWr Intervention — All participants will be asked to complete a secure confidential online survey focusing on needs assessment.
  Participants in the T-POWr Intervention Arm will receive a client-centered case management consultation based on how the participant responds to the online survey. The T-POWr will refer participants to assistance services based on the needs assessment, including accessing general health care, health insurance, hormone replacement therapy, housing, mental health care, domestic violence care, substance use treatment, etc. Each resource is extensively vetted to assure a trans-friendly experience and will be tailored to each geographic area across the project enrollment sites. The study facilitates referrals for services but will not provide extensive and ongoing case management.
  Arms: T-POWr Intervention Arm

SUMMARY:
CCTG 602 is a multisite demonstration project to evaluate the effectiveness of facilitated linkage to PrEP using a community-based transgender PrEP outreach worker (T-POWr) versus standard of care (SOC).

DETAILED DESCRIPTION:
Up to 500 self-identified transgender / gender non-conforming persons seeking daily Pre-Exposure Prophylaxis (PrEP) for the prevention of HIV will be enrolled into this study. Each participant will be followed up to 28 weeks after enrollment. The primary endpoint, successful linkage to a PrEP evaluation visit, will be measured after 30 days of enrollment.

Participants expressing interest in PrEP will be referred to the regional transgender PrEP outreach work (T-POWr) via phone call. Enrolled participants will be randomized (1:1) to either SOC PrEP linkage vs T-POWr facilitated PrEP linkage. Participants randomized into the SOC Arm will receive an HIV risk assessment, PrEP education, and an appointment for a linkage visit. Participants randomized into the T-POWr arm will receive SOC and a thorough client-centered case management evaluation that will assess needs including access to health insurance, general health care, assessment of current hormone administration, housing, mental health care, domestic violence care, substance use treatment, and other services.

Participants will be contacted at Week 4 to verify linkage, and at Weeks 16 and 28 to assess PrEP and HIV status, and access to referred services.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Self-identifies as a transgender or gender non-conforming person
* Self-identifies as HIV-negative or unknown status
* Ability to provide informed consent
* English or Spanish speaking

Exclusion Criteria:

* Severe active substance abuse or mental illness that the investigator feels will interfere with the ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender or Gender Non-conforming, defined as identifying with a gender different from sex assigned at birth.
Enrollment: 202 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Facilitated Linkage | Baseline up to Week 28
  To evaluate the effectiveness of a T-POWr intervention to effectively link transgender / gender non-conforming persons to a PrEP evaluation visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Morris, MD MPH, Study Chair — CCTG, UCSD AVRC
Locations (2):
- United States (2):
  - Los Angeles Lesbian, Gay, Bisexual, and Transgender Center, Los Angeles, California
  - UC San Diego AntiViral Research Center (AVRC), San Diego, California

IPD SHARING:
Plan to Share IPD: No